CLINICAL TRIAL: NCT05954065
Title: An Evaluation of the Effect of the Erchonia Corporation CFL Laser for Non-invasive Reduction of Submental Fat
Brief Title: An Evaluation of the Effect of the Erchonia Laser for Non-invasive Reduction of Submental Fat
Status: Completed | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-CHIN
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Erchonia CFL Laser (Experimental): 405nm violet and 520nm green laser light therapy.
  Interventions: Device: Erchonia CFL Laser

INTERVENTIONS:
Device: Erchonia CFL Laser — 405nm violet and 520nm green laser light therapy.

SUMMARY:
The purpose of this clinical study is to determine the effectiveness of the Erchonia® CFL (manufactured by Erchonia Corporation (the Company), in providing noninvasive fat reduction in the submental area.

DETAILED DESCRIPTION:
This clinical study is a prospective open-label design with post-study independent blinded outcome analysis to evaluate the efficacy of the Erchonia® CFL Laser in providing a noninvasive fat reduction in the submental area. Participants will receive 8 treatments over the course of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 65 years of age, inclusive.
* Submental and submandibular skin fold thickness > 1cm (measured by caliper).
* Subject agrees to maintain his/her weight (i.e., within 5%) by not making any major changes in diet or exercise routine during the course of the study.
* Subject agrees to abstain from partaking in any treatment to promote body contouring and/or weight loss during the course of study participation. Such treatments include, but are not limited to:

  * over-the-counter and/or prescription medications; dietary/herbal supplements and appetite suppressants.
  * weight loss programs/diet plans.
  * surgical procedures for sculpting of the chin fat pad/weight loss, e.g. submental lipectomy, lap bands.
* Subject has signed a written informed consent form.

Exclusion Criteria:

* Evidence of any cause of enlargement in the submental area other than localized subcutaneous fat, such as swollen lymph nodes or ptotic submandibular glands.
* Treatment with dermal fillers, radiofrequency or laser procedures, or chemical peels in the neck or chin area (below the mandible) within the past 6 months.
* Botulinum toxin or other aesthetic drug injections within the neck or chin area (below the mandible) within the past 6 months.
* History of a fat reduction procedure (e.g., liposuction, surgery, lipolytic agents, etc.) or implant in or adjacent to the area of intended treatment.
* Any dermatological conditions, such as scars in the location of the treatment area that may interfere with the treatment or evaluation.
* Active implanted device such as a pacemaker, defibrillator, or drug delivery system.
* Pregnant or intending to become pregnant in the next 6 months.
* Currently enrolled in a clinical study of an unapproved investigational drug or device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Glow Sculpting Spa, Harvey, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia CFL Laser
Started | 31
Completed | 30
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Erchonia CFL Laser
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.55 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 64.6 (3.03)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Accurately Identified Subject Pre- and Post-treatment Photographs by at Least Two of the Three Blinded Independent Evaluators.
Description: Reviewers will be blinded to post-treatment (12 weeks post) vs. baseline untreated area. The order in which images will be presented will be randomized. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. Success is defined as at least 2 of the 3 blinded evaluators correctly identifying a subject's pre-treatment and post-treatment (study endpoint) photographs for 80% or more of subjects.
Time Frame: 16 weeks (12 weeks post treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Erchonia CFL Laser
Number analyzed (Participants) | 30
Participants | 26

2. Secondary Outcome: Change in Submental Skinfold Thickness (mm)
Description: Submental skinfold thickness was measured using a standardized caliper technique applied consistently across all sites. The measurement involved pinching the submental tissue within the treatment area to capture a vertical skinfold, and recording the caliper reading in millimeters (mm). Because this technique folds the tissue, effectively doubling the fat layer thickness, the recorded value was divided by two to estimate the thickness of a single fat layer. This adjusted value was documented as the submental skinfold thickness (mm).
Time Frame: Baseline and 16 weeks (12 weeks post)
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Erchonia CFL Laser
Number analyzed (Participants) | 30
millimeters (mm) | -2.71 (1.12)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Erchonia CFL Laser
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT05954065/Prot_SAP_000.pdf